CLINICAL TRIAL: NCT05981222
Title: Biomechanical-matched Titanium Cages(Osteo Match) Versus PEEK Cages in Osteoporotic Lumbar Spine: a Multicenter, Prospective Cohort Study
Brief Title: Osteo Match Cages Versus PEEK Cages in Osteoporotic Patients
Acronym: OMC
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-397-04
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis; Degenerative Lumbar Disease; Degeneration Spine
Keywords: Osteoporosis; Cage subsidence; Lumbar fusion; Osteo Match
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Osteo Match cage: Patients undergoing posterior lumbar interbody fusion with Osteo Match Cages
- Peek Cage: Patients undergoing posterior lumbar interbody fusion with PEEK Cages

SUMMARY:
This is a multicenter, prospective cohort study. The osteoporotic patients requiring posterior lumbar interbody fusion(LIF) with cages are prospectively enrolled and followed up. The patients undergoing LIF with the biomechanical-matched 3D-printed titanium cages (Osteo Match) are compared with those using routine PEEK cages. The hypothesis is that the use of Osteo Match cages can reduce the rate of cage subsidence and increase the rate of lumbar fusion in osteoporotic patients.

DETAILED DESCRIPTION:
Interbody fusion cages are widely used for the surgical treatment of degenerative lumbar diseases, which can stabilize the spine and promote solid fusion. However, because of population aging and the high rate of osteoporosis in the elderly with lumbar degenerative diseases, the cage subsidence and failure of fusion have been frequently reported. The biomechanical strength (such as elasticity modulus) of routine PEEK cages is mismatched with osteoporotic bone, leading to cage subsidence and nonunion.

The 3D-printed porous titanium alloy cages have been proved to have advantages in speeding up and enhancing the lumbar fusion over conventional PEEK cages. However, most of the titanium cages still have much higher biomechanical strength than the osteoporotic bone. The new titanium cages named Osteo Match has been first clinically used in Peking University Third Hospital in China. The elastic modulus of Osteo Match cage is matched with that of lumbar spine with different degrees of osteoporosis. Therefore, we hypothesize that patients undergoing LIF with Osteo Match cages can achieve lower rate of cage subsidence and higher rate of lumbar fusion than those using PEEK cages.

The osteoporotic patients requiring posterior lumbar interbody fusion with cages are prospectively enrolled and followed up. The researchers will invite appropriate patients to participate in the study after their surgical plans are determined. General patients data are collected after informed consent, such as age, gender, weight, height, bone mineral density (measured by DXA, CT Hounsfield units, or QCT), detailed surgical plans, and etc. They are followed up at 3, 6, 12, and 24 months according to our clinical routine, including lumbar x-ray, CTand certain questions about the clinical outcomes.

The patients used Osteo Match cages are compared with those using conventional PEEK cages. The primary endpoints are the subsidence rate and fusion rate at 6 months follow-up. The secondary endpoints are the subsidence rate and fusion rate at other time point of follow-up , and the clinical outcomes(ODI/JOA/VAS) at every follow-up.

ELIGIBILITY:
Inclusion Criteria:

* aged≥ 50 years old
* lumbar degenerative diseases requiring lumbar fusion with pedicle screw fixation, such as degenerative lumbar spinal stenosis, degenerative lumbar spondylolisthesis.
* no response to nonoperative treatment of at least 3 months
* osteoporosis diagnosed by any method for bone mineral density evaluation, such as DXA, QCTor CT Hounsfield units
* requiring lumbar interbody fusion with cages within L3-S1
* the type of fusion cage has been chosen by the patients
* informed consent

Exclusion Criteria:

* the surgical plan includes any unconventional techniques used to strengthen the fixation, such as augmentation of the pedicle screw with bone cement
* lumbar spondylolisthesis of ≥II degree
* lumbar scoliosis of >20° or imbalance of spinal alignment
* history of lumbar fusion surgery
* cervical myelopathy, thoracic spinal stenosis, motor neuron disease,tuberculosis of spine,spinal tumor
* vertebral fracture within interbody fusion segement
* ASA of ≥IV

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The osteoporotic patients requiring lumbar interbody fusion with cages for lumbar degenerative diseases are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Cage subsidence rate | 6 months
  The presence of cage subsidence > 2mm at x-ray or CT images.
Fusion rate | 6 months
  The presence of continuous fusion mass at bone graft site in CT scans and absence of intervertebral mobility on lateral flextion-extension x-ray images.

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zou D, Yue L, Fan Z, Zhao Y, Leng H, Sun Z, Li W. Biomechanical Analysis of Lumbar Interbody Fusion Cages With Various Elastic Moduli in Osteoporotic and Non-osteoporotic Lumbar Spine: A Finite Element Analysis. Global Spine J. 2024 Sep;14(7):2053-2061. doi: 10.1177/21925682231166612. Epub 2023 May 3. PMID 37132375
- [Background] McGilvray KC, Easley J, Seim HB, Regan D, Berven SH, Hsu WK, Mroz TE, Puttlitz CM. Bony ingrowth potential of 3D-printed porous titanium alloy: a direct comparison of interbody cage materials in an in vivo ovine lumbar fusion model. Spine J. 2018 Jul;18(7):1250-1260. doi: 10.1016/j.spinee.2018.02.018. Epub 2018 Feb 26. PMID 29496624
- [Background] Li P, Jiang W, Yan J, Hu K, Han Z, Wang B, Zhao Y, Cui G, Wang Z, Mao K, Wang Y, Cui F. A novel 3D printed cage with microporous structure and in vivo fusion function. J Biomed Mater Res A. 2019 Jul;107(7):1386-1392. doi: 10.1002/jbm.a.36652. Epub 2019 Mar 18. PMID 30724479
- [Background] Goldstein CL, Brodke DS, Choma TJ. Surgical Management of Spinal Conditions in the Elderly Osteoporotic Spine. Neurosurgery. 2015 Oct;77 Suppl 4:S98-107. doi: 10.1227/NEU.0000000000000948. PMID 26378363
- [Background] Zou D, Jiang S, Zhou S, Sun Z, Zhong W, Du G, Li W. Prevalence of Osteoporosis in Patients Undergoing Lumbar Fusion for Lumbar Degenerative Diseases: A Combination of DXA and Hounsfield Units. Spine (Phila Pa 1976). 2020 Apr 1;45(7):E406-E410. doi: 10.1097/BRS.0000000000003284. PMID 31725127